CLINICAL TRIAL: NCT00941018
Title: A Randomized, Double Blind, Placebo Controlled, Ascending Single and Multiple Dose, Safety, Tolerability, Pharmacokinetic, Pharmacodynamic and Food Effect Study of RX-10001 in Healthy Volunteers
Brief Title: Single and Multiple Ascending Oral Dose Study of RX-10001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Resolvyx Pharmaceuticals, Inc (Industry)
Responsible Party: Per Gjorstrup, MD PhD Chief Medical Officier, Resolvyx
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RX-10001-002
Record Dates: First submitted 2009-07-14; First posted 2009-07-17 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Resolvins; RvE1; Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- SAD cohort 1 (Experimental): Single ascending dose (SAD) cohort 1 will participate in three dosing periods separated by 2 weeks. Eight subjects will be enrolled, 6 will receive RX-10001 and 2 will receive vehicle control. The starting dose will be 300 mg. Subsequent doses will be determined by the pk and safety data from previous cohorts.
  Interventions: Drug: RX-10001
- SAD cohort 2 (Experimental): SAD cohort 2 will participate in three dosing periods separated by 2 weeks. Eight subjects will be enrolled, 6 will receive RX-10001 and 2 will receive vehicle control. The doses to be administered will be determined by the pk and safety data from previous cohorts.
  Interventions: Drug: RX-10001
- MAD cohort 1 (Experimental): Multiple ascending dose (MAD) cohort 1 will consist of 10 subjects, 8 will receive RX-10001 and 2 will receive vehicle control. The dose of RX-10001 to be administered will depend upon the pk and safety results of the previous SAD cohorts.
  Interventions: Drug: RX-10001
- MAD cohort 2 (Experimental): MAD cohort 2 will consist of 10 subjects, 8 will receive RX-10001 and 2 will receive vehicle control. The dose of RX-10001 to be administered will depend upon the pk and safety results of the previous cohort.
  Interventions: Drug: RX-10001
- MAD cohort 3 (Experimental): MAD cohort 3 will consist of 10 subjects, 8 will receive RX-10001 and 2 will receive vehicle control. The dose of RX-10001 to be administered will depend upon the pk and safety results of the previous cohorts.
  Interventions: Drug: RX-10001
- MAD cohort 4 (Experimental): MAD cohort 4 will consist of 10 subjects, 8 will receive RX-10001 and 2 will receive vehicle control. The dose of RX-10001 to be administered will depend upon the pk and safety results of the previous cohort.
  Interventions: Drug: RX-10001

INTERVENTIONS:
Drug: RX-10001 — RX-10001 or vehicle control will be administered as an oral solution. Doses will be determined according to the pk results of the preceding cohorts.

SUMMARY:
This study is being conducted to determine the safety, tolerability, pharmacodynamics and pharmacokinetics of RX-10001.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18 - 32 kg/m2, inclusive
* Female subjects: must be of non-childbearing potential (either surgically sterilized or at least 1 year post-menopausal (amenorrhea duration of 12 months)
* Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "power drinks") and grapefruit (juice) from 48 h prior to entry in the clinical research center until discharge
* Medical history without major pathology
* Resting supine blood pressure and pulse rate showing no clinically relevant deviations as judged by the MI
* Computerised (12-lead) ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the MI
* All values for hematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the MI
* Willingness to sign the written Informed Consent Form (ICF)

Exclusion Criteria:

* Evidence of clinically relevant pathology
* Mental handicap
* History of relevant drug and/or food allergies
* Regular/routine treatment with non-topical medications within 30 days prior to drug administration
* Use of tobacco products (less than 60 days prior to drug administration)
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
* Use of concomitant medication (including over the counter medication, health supplements, multivitamins and vitamin C, vitamin and omega-3 supplements, and herbal remedies such as St. John's Wort extract) must have been stopped at least 14 days prior to the first dose. The use of a limited amount of acetaminophen (paracetamol) is permitted on discretion of the MI.
* Participation in a drug study within 60 days prior to drug administration. Participation in more than 3 other drug studies in the 10 months preceding the start of this study.
* Donation of more than 100 mL of blood within 60 days prior to drug administration. Donation of more than 1.5 litres of blood in the 10 months preceding the start of this study.
* Positive screen on drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids), barbiturates, benzodiazepines, tricyclic antidepressants and alcohol
* Intake of more than 24 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
* Positive screen on HBsAg
* Positive screen on anti HCV
* Positive screen on anti HIV 1/2
* Illness within 5 days prior to (the first) drug administration
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)), during work or during participation in a medical trial in the previous year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability following single and multiple ascending oral doses as assessed by adverse events, vital signs, 12-lead ECG, clinical laboratory and physical exam. | 1 and 7 days

SECONDARY OUTCOMES:
To determine the pk and pharmacodynamics after single and multiple ascending doses | 1 and 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Renger Tiessen, MD PhD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA International, Zuidlaren, Netherlands